CLINICAL TRIAL: NCT06618235
Title: A Phase I/IIa, Open-label, Dose Finding, Safety, Tolerability and Exploratory Trial of THEO-260 in Patients With High Grade Serous or Endometrioid Ovarian Cancer
Brief Title: Trial of THEO-260 in Ovarian Cancer Patients
Acronym: OCTOPOD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Theolytics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THEO-260-001
Record Dates: First submitted 2024-07-03; First posted 2024-10-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- THEO-260 (Experimental)
  Interventions: Biological: THEO-260

INTERVENTIONS:
Biological: THEO-260 — Oncolytic Virus

SUMMARY:
The goal of this clinical trial is to establish if THEO-260 is safe to administer to adult females with ovarian cancer. It will also aim to establish if THEO-260 is able to treat ovarian cancer. The main questions it aims to answer are:

* What medical problems do participants have when taking THEO-260?
* At what dose is THEO-260 both safe but also shows signs of being able to treat ovarian cancer?
* At the selected dose, test THEO-260 is a wider group of participants to confirm the safety and ability to treat ovarian cancer.

Part A will be the dose escalation/ finding part of the trial where we will aim to establish a Recommended Phase 2 Dose (RP2D).

Part B will be where the recommended RP2D is given to a larger group of participants.

Participants will:

* Be administered 6 doses of THEO-260 over the course of 2 weeks.
* They will then visit the clinic at regular intervals for check-ups and tests to monitor safety and THEO-260 ability to treat ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histological diagnosis of advanced high grade serous or endometrioid cancer of the fallopian tube, primary peritoneum or ovary either on archival biopsy or fresh tumour biopsy.
* Voluntary, written informed consent prior to trial procedures. Willingness and ability to comply with the protocol.
* Life expectancy of > 3 months.
* Adequate haematological and organ function (parameters apply).
* Non-pregnant and non-lactating and surgically sterile, or post-menopausal or abstinent or if of child-bearing potential will to use a highly effective form of contraception - where applicable.
* ECOG performance status of 0 or 1.
* Measurable disease as per RECIST V1.1.
* Part A: Platinum-resistant disease (radiological recurrence/ progression with 6 months of prior platinum treatment), primary platinum-refractory disease (recurrence/ progression during first line platinum treatment) and patients who are intolerant to or have no available SOC or SOC unacceptable/ unsuitable in the view of the Investigator. Part B: Advanced platinum-resistant disease: platinum-resistance as radiological recurrence/ progression within 6 months of prior platinum treatment or progression on SOC treatment or in intolerant to or has no available SOC or SOC unacceptable/ unsuitable in the view of the Investigator.

Exclusion Criteria:

* Prior anti-cancer treatment with 28 days or 5 half-lives whichever is longer, prior to first dose of THEO-260 or patients with unresolved or unstable serious toxic side-effects of prior chemotherapy or radiotherapy.
* Prior treatment with a group B adenovirus.
* Currently enrolled in a clinical trial of an IMP or used any IMP with 5 half-live, prior to first dose of THEO-260.
* Radiation therapy with 2 weeks of first dose of THEO-260 and is scheduled to have radiation therapy during participation of trial. Short courses of palliative radiation therapy should be discussed with the Medical Monitor and Sponsor.
* Clinical evidence of cerebral metastases or Central Nervous System (CNS) involvement including leptomeningeal disease. Patients with previous cerebral metastases must have no evidence of progression or haemorrhage after treatment and have been off dexamethasone for 4 weeks prior to first dose of THEO-260 with no ongoing requirement for dexamethasone or anti-epileptic drugs. Brain imaging in patients with a history of cerebral metastases or CNS involvement must not be older than 12 weeks (at the start of screening). Results of any unexpected or abnormal findings of brain imaging should be discussed with the Medical Monitor and Sponsor as part of the screening process.
* Uncontrolled pleural effusion or pericardial effusion requiring recurrent drainage procedures (as defined as once monthly or more frequently).
* Prior pneumonitis or history of interstitial lung disease.
* Confirmed QTcF ≥470 ms on screening 12-lead ECG or history of Torsades de pointes or history of congenital long QT syndrome.
* Concomitant medications that prolong the QTc interval and/or increase the risk for Torsades de Pointes that cannot be discontinued or substituted (within 5 half-lives or 14 days prior to the first dose of IMP, whichever was longer) with another drug prior to administration of IMP.
* Any other concurrent severe and/or uncontrolled medical or surgical condition which, in the view of the Investigator, could compromise the patient's participation in the trial due to safety, compliance concerns or ability to evaluate response.
* Patients with active hepatitis infection or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection. Patients positive for hepatitis C virus (HCV) antibodies are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Active infection with tuberculosis. Past or resolved tuberculosis is acceptable.
* Active infection with severe acute respiratory syndrome coronavirus 2 (SARS-Cov-2). All patients should be tested for active SARS-Cov-2 infection and have a negative COVID-19 result within 3 days of Day 1 (e.g., if a patient tested positive in antigen testing but asymptomatic, the patient will need to be excluded). Active infection with SARS-Cov-2 confirmed as per site's standard way of testing.
* Patients with active human immunodeficiency virus (HIV) infection or known history of HIV infection.
* Active infection requiring IV antibiotics within 2 weeks prior to first dose of THEO-260, or long-term oral therapy for systemic infection.
* Known contra-indications or hypersensitivity to the excipients of the IMP.
* Viral infection during the 2 weeks prior to first dose of THEO-260.
* Conditions requiring treatment with immunosuppressant medications or corticosteroids (except for patients receiving inhaled corticosteroids at a stable dose for a diagnosis of asthma) within 4 weeks prior to the first dose of THEO-260. Patients with steroid replacement due to immune-induced adrenal insufficiency would be eligible.
* Known risk of renal injury, including those with a past history of acute or sub-acute renal disease.
* Known heart failure New York Heart Association (NYHA) Class 2-4.
* Any major surgical procedure (planned or anticipated) (in the Investigator's judgement) within 2 weeks of the first dose of THEO-260 or within the anticipated treatment period.
* Known contra-indications or hypersensitivity to the AxMP, paracetamol.
* Known alcohol consumption in excess of 2 units per day.
* Part B: Greater than a single line of anti-cancer therapy in the platinum-resistant setting. Prior treatment with paclitaxel (either alone or in combination with Bevacizumab) in the platinum-resistant setting is allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of THEO-260 | Until end of trial for a participant, estimated at 1 year
  Safety and tolerability will be assessed by:
  Evaluation of DLTs and AEs during treatment and follow-up using National Cancer Institute (NCI) Common Terminology Criteria for AEs (CTCAE) v5.0 or American Society of Clinical Oncology (ASCO; for pneumonitis only) or American Society for Transplantation and Cellular Therapy (ASTCT; for cytokine release syndrome [CRS] only).
Establish recommended Phase 2 dose (RP2D) for THEO-260 | Until end of Part A of trial, estimated at 18 months after start of enrolment
  The totality of safety and efficacy data collected will be used to assess RP2D.
Evaluate preliminary efficacy of THEO-260 | Until end of trial, estimated at 3 years after start of enrolment
  The response to RP2D dose of THEO-260 will be assessed by Overall Response Rate (ORR) determined by tumour imaging according to RECIST v1.1.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of THEO-260 | Until Day 29 after first dose
  Assess PK profile (maximum concentration - Cmax) of THEO-260 in blood by qPCR.
Shedding of THEO-260 in saliva, urine and faeces | Until Day 29 after first dose
  Assess shedding of THEO-260 in buccal, urine and faecal samples by qPCR.
Risk of systemic cytokine release syndrome (CRS) after THEO-260 | Until Day 29 after first dose
  Assess systemic CRS following administration of THEO-260 by measurement of key markers in blood.
Evaluate preliminary efficacy of THEO-260 - RECIST | Until end of trial, estimated at 3 years after start of enrolment
  Determine response to THEO-260 as assessed by tumour imaging according to RECIST v1.1.
Evaluate preliminary efficacy of THEO-260 - CA125 | Until end of trial, estimated at 3 years after start of enrolment
  Efficacy will also be measured by changes in cancer antigen 125 (CA-125).

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - The Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Imperial College Healthcare NHS Trust, Hammersmith Hospital, London
  - Oxford University Hospitals NHS Foundation Trust, Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No